CLINICAL TRIAL: NCT04735575
Title: A First-in-human, Phase I/II, Open-Label Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Preliminary Antitumor Activity of EMB-06 in Patients With Relapsed or Refractory Multiple Myeloma
Brief Title: A Ph1/2 Study of EMB-06 in Participants With Relapsed or Refractory Myeloma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Company's resource optimization and product's development change
Sponsor: Shanghai EpimAb Biotherapeutics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EMB06X101
Record Dates: First submitted 2021-01-28; First posted 2021-02-03 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Relapsed or Refractory Multiple Myeloma
Keywords: Phase I/II; Bispecific antibody; BCMA; CD3; EMB-06; Immuno-oncology; Dose escalation; Cohort expansion; Relapsed or Refractory Multiple Myeloma; Hematological malignancy
MeSH Terms: conditions — Recurrence; Multiple Myeloma; Hematologic Neoplasms

STUDY DESIGN:
Intervention Model Description: Dose escalation followed by Cohort Expansion Phase at the RP2D.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- EMB-06 (Experimental): In Phase I part: participants enrolled at different time will receive EMB-06 by IV infusion at different ascending dose levels.
  In Phase II part: participants will receive EMB-06 by IV infusion at previously defined RP2D.
  Interventions: Biological: EMB-06

INTERVENTIONS:
Biological: EMB-06 — EMB-06 is a FIT-Ig® bispecific antibody against BCMA and CD3.

SUMMARY:
The primary purpose of this study is to identify the recommended Phase 2 dose(s) (RP2Ds) and schedule assessed to be safe for EMB-06 and to characterize the safety and tolerability of EMB-06 at the RP2Ds. Pharmacokinetics (PK), immunogenicity, and the anti-multiple myeloma activity of EMB-06 will also be assessed.

DETAILED DESCRIPTION:
This is a Phase I/II, multi-center, open label, multiple-dose, first in human study, designed to assess safety and tolerability, and to identify the maximum tolerated dose (MTD) and/or recommended Phase 2 dose (RP2D) for EMB-06 in patients with relapsed or refractory multiple myeloma. Pharmacokinetics, pharmacodynamics, immunogenicity, and response will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand and willing to sign the informed consent form (ICF)
* Patients who have been diagnosed with multiple myeloma according to IMWG diagnostic criteria 2014 and have relapsed or refractory multiple myeloma with at least one measurable lesion.
* The patient must have received at least two lines (for patients in the US, at least three lines which should include anti-CD38 antibody) of prior antimyeloma therapies, and must have received treatment with proteasome inhibitors, immunomodulatory agents, and if accessible, an anti-CD38 targeting monoclonal antibody.
* ECOG performance status 0 or 1 for phase I, and ≤2 for phase II.
* Adequate organ function and reasonable laboratory test results to participate in the trial.
* Highly effective contraception

Exclusion Criteria:

* Life expectancy is less than 3 months.
* Patient participated in any other clinical study within 1 month prior to enrollment in this clinical study.
* Patients with ongoing AE.
* Previously treated with any BCMA-targeted therapy.(Exception: in Phase 2 portion, up to 10 patients who have received prior anti-BCMA ADC or BCMA targeted CAR-T can be enrolled)
* History of allogeneic stem cell transplantation.
* Previously treated with the following anti-tumor therapy (prior to first dosing of EMB-06)

  1. Treated with monoclonal antibody for multiple myeloma within 28 days
  2. Treated with proteasome inhibitors within 14 days
  3. Treated with immunomodulatory agents within 14 days
  4. Treated with cytotoxic therapy within 14 days
  5. Received investigational drug within 28 days or at least 5 half-lives, whichever is shorter (if a, b, c, d not applicable)
  6. Received radiotherapy within 21 days. Except that the radiation portal covered ≤ 5% of the bone marrow reserve, the patient will be eligible to participate in the study regardless of the end date of radiation therapy
  7. Plasmapheresis within 7 days
* Patient received autologous stem cell transplantation within 12 weeks prior to the start of study treatment.
* Active or historically multiple myeloma related central nervous system involvement.
* Patients requiring high dose of systemic treatment with corticosteroids.
* Patients with active infections, including COVID-19, hepatitis, etc..
* History of severe allergic reactions
* Patients with severe or uncontrolled cardiovascular disorder requiring treatment
* Pre-existing other serious medical conditions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-05-20 (Actual); Primary Completion 2024-08-20 (Actual); Study Completion 2024-08-20 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of adverse events | Screening up to follow-up (30 days after the last dose)
  Incidence and severity of AE.
Incidence of serious adverse events (SAE) | Screening up to follow-up (30 days after the last dose)
  Incidence of SAE
Incidence of dose interruptions. | Screening up to follow-up (30 days after the last dose)
  Incidence of dose interruptions of EMB-06 during treatment as a measure of tolerability.
Dose intensity | Screening up to follow-up (30 days after the last dose)
  Actual amount of drug taken by patients divided by the planned amount.
The incidence of DLTs during treatment. | First infusion to the end of Cycle 1 (each cycle is 28 days)
  The Dose Limiting Toxicities (DLTs) are based on drug related adverse events and are specifically defined in study protocol.
Overall Response Rate (ORR) | From the date of dosing until the date of first documented progression or date of death from any cause, whichever came first, expected average 6 months
  Measured by IMWG criteria, only applicable in Phase II part

SECONDARY OUTCOMES:
Area under the serum concentration-time curve (AUC) of EMB-06. | Through treatment until EOT visit, expected average 6 months
  Blood samples for serum PK analysis will be obtained (AUC).
Maximum serum concentration (Cmax) of EMB-06. | Through treatment until EOT visit, expected average 6 months
  Blood samples for serum PK analysis will be obtained (Cmax).
Trough concentration (Ctrough) of EMB-06. | Through treatment until EOT visit, expected average 6 months
  Blood samples for serum PK analysis will be obtained (Ctrough).
Average concentration over a dosing interval (Css, avg) of EMB-06. | Through treatment until EOT visit, expected average 6 months
  Blood samples for serum PK analysis will be obtained (Css, avg).
Terminal half-life (T1/2) of EMB-06. | Through treatment until EOT visit, expected average 6 months
  Blood samples for serum PK analysis will be obtained (T1/2).
Systemic clearance (CL) of EMB-06. | Through treatment until EOT visit, expected average 6 months
  Blood samples for serum PK analysis will be obtained (CL).
Steady state volume of distribution (Vss) of EMB-06. | Through treatment until EOT visit, expected average 6 months
  Blood samples for serum PK analysis will be obtained (Vss).
Progression free survival (PFS) of EMB-06 as assessed by IMWG criteria. | From the date of dosing until the date of first documented progression or date of death from any cause, whichever came first, expected average 6 months
  Preliminary anti-multiple myeloma activity of EMB-06 will be obtained (PFS).
Duration of response of EMB-06 as assessed by IMWG criteria | From the date of dosing until the date of first documented progression or date of death from any cause, whichever came first, expected average 6 months
  Preliminary anti-multiple myeloma activity of EMB-06 will be obtained (DOR).
Incidence and titer of anti-drug antibodies stimulated by EMB-06. | Up to End of Treatment Follow Up Period (30 days after the last dose)
  Antibodies to EMB-06 will be assessed to evaluate potential immunogenicity.

CONTACTS AND LOCATIONS:
Locations (10):
- Australia (3):
  - Sunshine Coast Haematology and Oncology Clinic (SCHOC), Buderim, Queensland
  - Epworth Healthcare, Richmond, Victoria
  - One Clinical Research (OCR), Nedlands, Western Australia
- China (7):
  - Beijing Jishuitan Hospital, Beijing, Beijing Municipality
  - Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Peking University, Third Hospital, Beijing
  - Guangdong Provincial People's Hospital, Guangzhou
  - The First Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou
  - Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan
  - Henan Cancer Hospital, Zhengzhou

IPD SHARING:
Plan to Share IPD: No